CLINICAL TRIAL: NCT03866824
Title: MENIPREP Study: Evauation of the Effectiveness of Prp Injection in the Management of Degenerative Meniscal Lesions : Randomized Controlled Trial Double Blind Versus Reference Treatment"
Acronym: MENIPREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-55; 2018-A02497-48 (Other: IDRCB)
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: DEGENERATIVE MENISCAL LESIONS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental)
  Interventions: Drug: injection of Platelet Enhanced Plasma(PRP); Device: RMI
- reference treatment (Active Comparator)
  Interventions: Drug: injection of corticosteroids; Device: RMI

INTERVENTIONS:
Drug: injection of Platelet Enhanced Plasma(PRP) — intra-articular injection
  Arms: PRP group
Drug: injection of corticosteroids — intra-articular injection
  Arms: reference treatment
Device: RMI — A CONTROL RMI at 1 year follow-up.

SUMMARY:
Meniscal tissue has very limited intrinsic properties in terms of repair, given the low mitotic activity of chondrocytes and poor vascularization. Nevertheless, its capacity for regeneration, in vivo and in vitro, can be stimulated by the contribution of growth factors, as has been widely described in the medical and scientific literature. Platelet Enhanced Plasma (PRP) is an autologous biological product (that is, derived from the patient's blood) containing a growth factor concentrate. The contribution of these growth factors stimulates cartilage repair by stimulating neovascularization, collagen synthesis and activation of chondrocytes. Intra-articular injection PRP is an autologous biological product, now used in daily practice for the treatment of early osteoarthritic lesions.

The hypothesis of this work is that the injection of PRP in contact with LMD(Degenerative Meniscal Lesions) will improve the clinical symptomatology of our patients compared to reference treatment (intra-auricular injection of corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 20 to 80

* MDD diagnosis objected to MRI (grade II/III)
* Joint pain for more than 3 month
* Absence of bone lesion or moderate knee osteoarthritis stage <2 on the Kellgren Laurence scale (objectified on radiography in schuss) in the 6 months prior to inclusion
* Axial deformity of the lower limbs less than or equal to 5 °
* Signed consent signed by the patient
* Ability to perform procedures as part of the follow-up (walk 50 steps on a flat surface and up / down stairs).
* Be affiliated to a health insurance scheme

Exclusion Criteria:

* Axial deformity> 5 °
* Ligament instability
* Major injuries or surgery of the target knee or lateral contralateral knee in the 12 months preceding the inclusion visit
* Ligament reconstruction in the 12 months prior to the inclusion visit
* Need a cane or assistance to move
* BMI> 35
* Thrombocytopenia <150 G / L
* Thrombocytosis> 450 G / L

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Control by Magnetic Resonance Imaging (MIR) | 12 Months
  To evaluate the evolution of the LMD compared to pretherapeutic images.

SECONDARY OUTCOMES:
self-completed questionnaire EVA score | 12 Months
  EVA (analogical visual scale)
self-completed questionnaire SF36 | 12 Months
  SF36 (The Short Form (36) Health Survey)
self-completed questionnaire KOOS score | 12 Months
  KOOS (Knee Injury and Osteoarthritis Outcome Score)

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France